CLINICAL TRIAL: NCT04133467
Title: The Scalp Block for Postoperative Pain Control in Craniosynostosis Surgery: a Case Control Study
Brief Title: Scalp Block Decreases Pain and Side Effects
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2024
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Craniosynostoses; Pain, Postoperative
MeSH Terms: conditions — Craniosynostoses; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group SB: Scalp block performed with Levobupivacaine 0.125% (total dose 2 mg/kg) in combination with intraoperative intravenous acetaminophen (15 mg/kg if body weight >10Kg, 7 mg/kg if body weight < 10 kg).
  Interventions: Other: scalp block
- Group ST: intravenous acetaminophen according to the body weight, plus intravenous tramadol 1 mg/kg

INTERVENTIONS:
Other: scalp block — intravenous acetaminophen according to the body weight, plus intravenous tramadol 1 mg/kg)
  Other Names: intravenous pharmacological approach
  Groups: Group SB

SUMMARY:
Postoperative analgesia after corrective surgery of paediatric craniosynostosis is crucial in term of short and long-term outcomes. The objective of this observational case- control study was to evaluate the effectiveness of an analgesic technique based on the scalp block versus traditional pharmacological approach.

DETAILED DESCRIPTION:
Several studies on craniosynostosis and the correlated risk factors have been published, the majority of them focusing on the perioperative management of blood losses and avoidance of haemorrhagic shock. Other issues related to anaesthetic management of the surgical correction of craniosynostosis are metabolic and electrolyte disturbances.

Even if craniosynostosis surgery is an invasive procedure, there is a current misconception that it would be associated with minimal pain, despite the extensive exhibition of the skull and periostea dissection. The Literature about the assessment and management of postoperative pain in this particular surgical setting is scarce. Assessment of pain in infants is challenging, and often relies on clinical observation. To date, there are no evaluative and therapeutic parameters globally accredited in this category of patients. The scalp nerve block (SNB) is a regional anaesthetic technique, performed since several years in children undergoing a variety of procedures, from neurosurgery to eye-nose-throat surgery.SNB has been proposed as a complement to the routine craniosynostosis anaesthetic protocol, and should be associated to a reduced need for opioids.

Thirteen patients, aged between 3 months and 2 years, undergoing cranioplasty for the correction of craniosynostosis were subjected to SNB (Group SB) with Levobupivacaine 0.125% (total dose 2 mg/kg), performed before awakening, in combination with intraoperative intravenous acetaminophen (15 mg/kg if body weight >10Kg, 7 mg/kg if body weight < 10 kg). The SNB procedure was performed using the modified Pinosky technique, with levobupivacaine 0,125%(10). A targeted infiltration of 0,75-2ml of local anaesthetic (LA) solution was done at multiple sites with a 23G needle.

This Group of patients were compared with another group of 13 patients, derived from our database, and treated with the traditional pharmacological approach given intraoperatively (intravenous acetaminophen according to the body weight, plus intravenous tramadol 1 mg/kg).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cranioplasty for the correction of craniosynostosis

Exclusion Criteria:

* allergies to local anesthetics and/or analgesics
* specific drug therapies (pain relievers, sedatives and/or epileptic)
* denied consent to the study; development of postoperative intracranical bleeding and/or gastrointestinal bleeding
* need of nasogastric tube
* development of gastrointestinal infections.

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with aged between 3 months and 2 years, undergoing cranioplasty for the correction of craniosynostosis
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | OPS was assessed until the fifth day of hospitalization.
  Objective Pain Score incorporates four pain behaviors (crying, movement, agitation, and verbalization) and was evaluated at following times:
  * 30 minutes after extubation (T0)
  * 2 hours after extubation (T1)
  * 4 hours after extubation (T2)
  * 8 hours after extubation (T3)
  * at discharge from Pediatric Intensive Care Unit (T4).
  * at in the Neurosurgical ward OPS was assessed every eight hours, until the fifth day of hospitalization.

SECONDARY OUTCOMES:
resumption of oral nutrition | first postoperative day
  evaluation of post-operative feeding recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Rossano festa, MD, Principal Investigator — Fondazione Universitaria Policlinico Gemelli IRCCS roma Italia
Locations (1):
- Rossano Festa, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stricker PA, Goobie SM, Cladis FP, Haberkern CM, Meier PM, Reddy SK, Nguyen TT, Cai L, Polansky M, Szmuk P, Fiadjoe J, Soneru C, Falcon R, Petersen T, Kowalczyk-Derderian C, Dalesio N, Budac S, Groenewald N, Rubens D, Thompson D, Watts R, Gentry K, Ivanova I, Hetmaniuk M, Hsieh V, Collins M, Wong K, Binstock W, Reid R, Poteet-Schwartz K, Gries H, Hall R, Koh J, Bannister C, Sung W, Jain R, Fernandez A, Tuite GF, Ruas E, Drozhinin O, Tetreault L, Muldowney B, Ricketts K, Fernandez P, Sohn L, Hajduk J, Taicher B, Burkhart J, Wright A, Kugler J, Barajas-DeLoa L, Gangadharan M, Busso V, Stallworth K, Staudt S, Labovsky KL, Glover CD, Huang H, Karlberg-Hippard H, Capehart S, Streckfus C, Nguyen KT, Manyang P, Martinez JL, Hansen JK, Levy HM, Brzenski A, Chiao F, Ingelmo P, Mujallid R, Olutoye OA, Syed T, Benzon H, Bosenberg A; Pediatric Craniofacial Collaborative Group. Perioperative Outcomes and Management in Pediatric Complex Cranial Vault Reconstruction: A Multicenter Study from the Pediatric Craniofacial Collaborative Group. Anesthesiology. 2017 Feb;126(2):276-287. doi: 10.1097/ALN.0000000000001481. PMID 27977460
- [Background] Thomas K, Hughes C, Johnson D, Das S. Anesthesia for surgery related to craniosynostosis: a review. Part 1. Paediatr Anaesth. 2012 Nov;22(11):1033-41. doi: 10.1111/j.1460-9592.2012.03927.x. PMID 22928738
- [Background] Chiaretti A, Pietrini D, Piastra M, Polidori G, Savioli A, Velardi F, Ciano F, Di Rocco C. Safety and efficacy of remifentanil in craniosynostosis repair in children less than 1 year old. Pediatr Neurosurg. 2000 Aug;33(2):83-8. doi: 10.1159/000028981. PMID 11070434
- [Background] Teo JH, Palmer GM, Davidson AJ. Post-craniotomy pain in a paediatric population. Anaesth Intensive Care. 2011 Jan;39(1):89-94. doi: 10.1177/0310057X1103900115. PMID 21375097
- [Background] Guilfoyle MR, Helmy A, Duane D, Hutchinson PJA. Regional scalp block for postcraniotomy analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 May;116(5):1093-1102. doi: 10.1213/ANE.0b013e3182863c22. Epub 2013 Mar 11. PMID 23477962
- [Background] Pinosky ML, Fishman RL, Reeves ST, Harvey SC, Patel S, Palesch Y, Dorman BH. The effect of bupivacaine skull block on the hemodynamic response to craniotomy. Anesth Analg. 1996 Dec;83(6):1256-61. doi: 10.1097/00000539-199612000-00022. PMID 8942596
- [Background] Pardey Bracho GF, Pereira de Souza Neto E, Grousson S, Mottolese C, Dailler F. Opioid consumption after levobupivacaine scalp nerve block for craniosynostosis surgery. Acta Anaesthesiol Taiwan. 2014 Jun;52(2):64-9. doi: 10.1016/j.aat.2014.05.006. Epub 2014 Jun 21. PMID 25016510
- [Background] Phillips S, Gift M, Gelot S, Duong M, Tapp H. Assessing the relationship between the level of pain control and patient satisfaction. J Pain Res. 2013 Sep 9;6:683-9. doi: 10.2147/JPR.S42262. eCollection 2013. PMID 24049457
- [Derived] Festa R, Tosi F, Pusateri A, Mensi S, Garra R, Mancino A, Frassanito P, Rossi M. The scalp block for postoperative pain control in craniosynostosis surgery: a case control study. Childs Nerv Syst. 2020 Dec;36(12):3063-3070. doi: 10.1007/s00381-020-04661-z. Epub 2020 May 17. PMID 32418049